CLINICAL TRIAL: NCT06043947
Title: Survival Monitoring in Russian Cancer Registries
Acronym: SURVIMON
Status: Active, not recruiting | Type: Observational
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Collaborators: European University at St. Petersburg (Other)
Responsible Party: Sponsor
Other Study IDs: SURVIMON-2023
Record Dates: First submitted 2023-09-11; First posted 2023-09-21 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Melanoma; Breast Cancer; Oncology; Colon Cancer; Prostate Cancer; Survivorship; Lung Cancer; Cervix Cancer
Keywords: Survivorship survey; Survivorship care; Oncology; Melanoma; Breast cancer; Lung cancer
MeSH Terms: conditions — Melanoma; Breast Neoplasms; Neoplasms; Colonic Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to establish a holistic framework for continuous cancer survival surveillance in Russian regions with high-quality population-based cancer registry data. The data from the population-based cancer registries of the Northwestern regions of Russia will be used to assess net and cause-specific survival trends.

DETAILED DESCRIPTION:
The main sources of cancer incidence data in Russia are population-based cancer registries (PBCR). National recommendations guide the content of corresponding variables stored in PBCRs. Data were collected for the following regions: Arkhangelsk Oblast and Nenets Autonomous Okrug (combined), Republic of Karelia, Komi Republic, Vologda Oblast, Kaliningrad Oblast, Leningrad Oblast, Murmansk Oblast, Novgorod Oblast, Pskov Oblast, and St. Petersburg. Quality assessment procedures will be applied to the population-based cancer registries (PBCRs) datasets. Essential variables will be extracted following the recommended list of ENCR/IACR.

The list of variables consists of two classes: original variables present in PBCRs datasets and synthetic variables calculated based on the original variables. "IARC/IACR Tools for Cancer Registries" (IARC tools) software was used for the data cleaning, conversion to ICD-O-3, and multiple primaries assessment. Duplicates were removed by applying IARC/IACR/ENCR multiple primary rules. The analysis is limited to twenty years: 2000 - 2021.

The Federal State Statistics Service (FSSS) is the primary regional and national mortality data source. However, the raw data from this source has several drawbacks. The main problem is the absence of the distribution of persons with undetermined ages and/or causes of death. The data sets for this research are obtained from the Russian Fertility and Mortality Database (RFMD) of the Center for Demographic Research of the New Economic School. The RFMD database is based on the FSSS data but has a higher data quality due to the redistribution of deaths with the abovementioned characteristics. This source's population and mortality data contained the following variables: region, year, sex, age (5-year age groups from 0 to 85+), and cause of death.

Population data was obtained from the same source. The data were based on the 1989, 2002 and 2010 population censuses. It has been extrapolated to other years using annual statistics on mortality and births.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of any age
* Data record meets IARC/IACR Tools for Cancer Registries requirements

Exclusion Criteria:

* Severe patient data missing from a record

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patient population, that were diagnosed and registered in regions covered by PBCR.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Net survival | From the date of diagnosis to the date of death (up to 10 years)
  Net survival computed using Pohar-Perme method.
Cause-specific survival | From the date of diagnosis to the date of death (up to 10 years)
  Rates calculated using Kaplan-Maier method.

CONTACTS AND LOCATIONS:
Locations (1):
- N. N. Petrov Research Institute of oncology, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barchuk A, Tursun-Zade R, Belayev A, Moore M, Komarov Y, Moshina N, Anttila A, Nevalainen J, Auvinen A, Ryzhov A, Znaor A. Comparability and validity of cancer registry data in the northwest of Russia. Acta Oncol. 2021 Oct;60(10):1264-1271. doi: 10.1080/0284186X.2021.1967443. Epub 2021 Aug 23. PMID 34424113